CLINICAL TRIAL: NCT00821756
Title: The Amager Project. Intervention After Suicide Attempt: A Randomized Study.
Brief Title: The Amager Project: Intervention After Suicide Attempt
Acronym: Amager
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Ministry of Social Affairs, Denmark (Other Government)
Responsible Party: August G. Wang, Psychiatric Centre Amager, Copenhagen, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AH-2005
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2009-01

CONDITIONS: Suicidal Behaviour; Repetition of Suicidal Behaviour
Keywords: Suicidal behaviour; Attempted suicide; Self harm; Suicide; Health system contacts; Contacts with health system
MeSH Terms: conditions — Suicide, Attempted; Self-Injurious Behavior; Suicide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Assertive intervention in OPAC-style: Outreach,problem solving,adherence,continuity
  Interventions: Behavioral: OPAC (Outreach, Problem solving, Adherence, Continuity)
- 2 (No Intervention): Control arm: Treatment as usual

INTERVENTIONS:
Behavioral: OPAC (Outreach, Problem solving, Adherence, Continuity) — Assertive outreach immediately after the suicide attempt with about 8 home visits plus contact by telephone, phone messages, e-mails. Duration of intervention 6 months.
  Arms: 1

SUMMARY:
Background:

Repetition rate after a suicide attempt and self harm is very high, about 12-30 percent. Studies, reviewed by Hawton, 1999 show a lack of evidence for psychosocial interventions. Compliance with aftercare is also often very poor.

Objective:

Inspired by the Norwegian Baerum project, the aim is to study if active, assertive outreach, seeking contact, talking about problem solution, motivate to comply to other appointments, will reduce repetition of suicidal acts in the following years.

Methods:

The design is a prospective randomized, controlled trial. The patients (immediately after a suicide attempt or deliberate self harm)) included are randomized to intervention or standard (treatment as usual), aiming at at least 60 persons in each arm. The intervention is carried out through research nurses with about 8 home visits, phone contact, phone messaging, e-mails.Included are persons 12 years of age and older, danish speaking without translator and without diagnoses of severe mental illness (schizophrenia, bipolar illness, mania and severe/psychotic depression) or severe dementia.

Results:

Outcome is measured by repetition of suicidal act (suicide attempt, self harm or completed suicide)as recorded in medical records and by the Danish Cause of Death Register. Repetition measured by persons and by acts throughout 1 year, 2 and 3 years periods. Additional outcome is number and character of health system contacts.

ELIGIBILITY:
Inclusion Criteria:

* Suicide attempt and self harm

Exclusion Criteria:

* Severe mental diagnosis (schizophrenia, psychosis, bipolar affective disorder, severe/psychotic depression, severe dementia)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2005-01; Primary Completion 2008-08 (Actual); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Persons repeating a suicidal act | One, two and three years

SECONDARY OUTCOMES:
Acts of suicidal behaviour Contacts with health system | One, two and three years

CONTACTS AND LOCATIONS:
Overall Officials: August G. Wang, M.D., Principal Investigator — Psychiatric Centre Amager, Copenhagen University Hospital
Locations (1):
- Psychiatric Centre Amager, Copenhagen University Hospital, Copenhagen S, Denmark

REFERENCES:
- [Background] Hvid M, Wang AG. Preventing repetition of attempted suicide--I. Feasibility (acceptability, adherence, and effectiveness) of a Baerum-model like aftercare. Nord J Psychiatry. 2009;63(2):148-53. doi: 10.1080/08039480802423022. PMID 19016074
- [Derived] Hvid M, Vangborg K, Sorensen HJ, Nielsen IK, Stenborg JM, Wang AG. Preventing repetition of attempted suicide--II. The Amager project, a randomized controlled trial. Nord J Psychiatry. 2011 Oct;65(5):292-8. doi: 10.3109/08039488.2010.544404. Epub 2010 Dec 20. PMID 21171837